CLINICAL TRIAL: NCT02025686
Title: Hyperbaric Oxygen Therapy Attenuates Central Sensitization Induced by a Thermal Injury in Human Volunteers (HBO)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Per Rotbøll Nielsen (Other)
Responsible Party: Sponsor-Investigator, Per Rotbøll Nielsen, Consultant, Rigshospitalet, Denmark
Organization: Rigshospitalet, Denmark (Other)
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Basic Science
Other Study IDs: HBO12-04-2013; 2011-41-6327 (Other: Danish Data Protection Agency)
Record Dates: First submitted 2013-12-09; First posted 2014-01-01 (Estimated); Last update posted 2014-01-01 (Estimated); Status verified 2013-12

CONDITIONS: Pain; Inflammation; Hyperalgesia
Keywords: Pain; Inflammation; Hyperalgesia; burn injury; Hyperbaric Oxygen
MeSH Terms: conditions — Pain; Inflammation; Hyperalgesia; Burns | interventions — Hyperbaric Oxygenation

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Hyperbaric Oxygen (Experimental): Subjects will breathe oxygen (FIO2 = 1.0) at 2.4 ATA in a hyperbaric chamber after the tonic heat stimulations. The duration of oxygen exposure is 90 min
  Interventions: Drug: Hyperbaric Oxygen; Other: Normal ambient conditions

INTERVENTIONS:
Drug: Hyperbaric Oxygen — Subjects will breathe oxygen (FIO2 = 1.0) at 2.4 ATA in a hyperbaric chamber after the tonic heat stimulations. The duration of oxygen exposure is 90 min.
Other: Normal ambient conditions — Normal ambient conditions (1 ATA, FIO2 = 0.21)

SUMMARY:
The hypothesis of this investigation is to observe if HBO have an anti-inflammatory effect in humans induced by tonic heat stimulation. It has been shown in animal studies with rats that HBO could reduce the paw edema induced by carrageenan as an inflammatory agent. The authors are not aware of similar studies in human subjects investigating this effect of HBO. Aim: To investigate the anti-inflammatory effect of HBO by reducing the hyperalgesia induced by heat stimulation in healthy subjects and promote future research and understanding of the anti-inflammatory processes in humans. The primary endpoint is a reduced area of secondary hyperalgesia after HBO.

ELIGIBILITY:
Inclusion Criteria:

* Age > 18 yr Approved physical health examination Healthy Male

Exclusion Criteria:

* Arterial hypertension Chronic pain Claustrophobic tendency History of substance abuse Impaired cognitive abilities Inability to participate in quantitative sensory testing Incomplete understanding of Danish Neurological deficits Previous barotrauma or pneumothorax Previous head trauma Unable to equilibrate pressure in middle ear and/or sinuses

Min Age: 18 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 16 (Actual)
Dates: Start 2012-03; Primary Completion 2012-08 (Actual); Study Completion 2012-10 (Actual)

PRIMARY OUTCOMES:
The effect of Hyperbaric Oxygen Therapy on Pain and Inflammation induced by Tonic Heat Stimulation in Human Volunteers | 8 weeks
  Inflammation

SECONDARY OUTCOMES:
Pain on Pain Scores on the Visual Analog Scale | 8 weeks

CONTACTS AND LOCATIONS:
Locations (1):
- Copenhagen University Hospital, Rigshospitalet, Copenhagen, Denmark